CLINICAL TRIAL: NCT05681832
Title: Developing a Physical Activity Program Based on Behavior Change Models in Children and Investigation of Its Efficiency.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Mira Amer, BSc.P.T., Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-74555795-050.01.04-567380
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Behavior, Child; Physical Inactivity
Keywords: child; behavior change models; HIIT; Exercise; physical activity; physical inactivity; motivation
MeSH Terms: conditions — Child Behavior; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Intervention group
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Intervention group — The children in this group will participate in a 15-minute HIIT (High-intensity interval training) program twice a week for eight weeks. Motivational interviewing through presentations and Kahoot for the children and their parents will be done at the program's beginning, middle, and end.
  The HIIT program will consist of 2.5 minutes of warm-up 12.5 exercises then a cool-down period of 5 minutes. The intensity of the exercise was increased based on each kid's performance and monitored during the sessions using a smartwatch.
  Arms: Intervention group

SUMMARY:
The aim of our study is to develop a physical activity program based on behavioral change models for children and to investigate the effectiveness of the physical activity program we have developed for children attending primary school. There is a limited number of studies in the literature on exercise habits in children, and there is no evidence on which model will provide better results when integrated into school or training programs. Although behavioral modification-based physical activity programs for children have been established and their effectiveness has been investigated in many different countries, there are limited randomized controlled studies on this subject. Currently, there are no randomized control studies on the topic in Turkey.

Our study will be the first study in which a school-based physical activity program based on behavioral change models in Turkish children is developed and its effectiveness is investigated. We believe that our study will contribute to the development of new models and protocols to improve the health of children in Turkey and the world and to provide behavior change methods that are research-based to combat physical inactivity.

DETAILED DESCRIPTION:
The COVID-19 pandemic, which started in 2019, has negatively affected the lives of all humanity in many ways, especially with the decrease in physical activity. Due to quarantines, schools continued their educational activities online for a long time. While physical inactivity in children was a serious problem even in the pre-pandemic period, the restrictions imposed due to pandemic conditions had a catastrophic effect on the physical inactivity levels of children. It has been reported that children reach the recommended physical activity levels while they are at school. Studies show that the habits we have acquired since childhood are most likely habits that we can have for a lifetime.

The effectiveness of behavior change theories and models has been proven in studies conducted to gain exercise habits in various age groups. In the literature, many theories such as Self-Determination Theory (SDT), Transtheoretical Model, Planned Behavior Theory, and Social Cognitive Theory have been used to help children gain exercise habits. In a cross-sectional study involving 462 children aged 7-11, the effectiveness of the SDT model on children's physical activity motivation was examined. The results showed that there is a positive relationship between children's motivation based on activity enjoyment and satisfaction and physical activity scores. It has been reported that applications based on theory are promising for future interventions aimed at increasing physical activity levels in children.

However, there is a limited number of studies in the literature to gain exercise habits in children, and there is no evidence that which model will provide better results. In a postgraduate thesis done in Turkey in 2021, online exercise training based on behavior change theories and strategies was applied to gain exercise habits in children. They reported limited evidence that they obtained Although very few children participated in the study due to restrictions during the COVID-19 pandemic, they reported limited evidence that children achieved positive changes in health behavior.

For these reasons, the planning of our study is to develop a physical activity program based on behavioral change models for children and to investigate the effectiveness of the physical activity program we have developed in children attending primary school.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily wanting to join the program
* Not having any chronic diseases
* Be able to read and write
* To have the cognitive skills to understand and answer the questionnaire
* To be a student at primary or secondary school.

Exclusion Criteria:

* Having a vision or hearing problem
* Have a diagnosis of chronic cardiac, neurological, or rheumatic disease
* Doing regular exercise/sports for the last 6 months

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
The Cognitive Behavioral Physical Activity Questionnaire | Change from baseline to 8 weeks
  This questionnaire will test the changes in behavior towards physical activity in children. The scale consists of 3 sub-dimensions, namely self-regulation and personal barriers, and a total of 15 statements. All statements in the scale are scored with a 5-point Likert Type rating as "1. I totally disagree,…, 5. I totally agree".
The physical Activity Stages Of Change Questionnaire | Change from baseline to 8 weeks
  This questionnaire will specifiy which stage of change the child is in according to the transtheoretical model. Transtheoretical Model, explains whether the individual is ready to change their behavior and describes the behavior change process that occurs in stages. This will help us know how to modify the program to work out well for each child.
Motivation Scale For Participation In Physical Activity | Change from baseline to 8 weeks
  This scale will evaluate the level of motivation to participate in physical activity.
The physical activity efficacy scale | Change from baseline to 8 weeks
  This scale consists of 5 dimensions and 26 items (at school: 6 items, transportation: 3 items, indoor: 5 items, leisure and recreation: 6 items, in-school travel and transportation: 6 items). The scale consists of two parts. In the first part, demographic information is asked, and in the second part, how much they trust themselves to take part in physical activities in the five physical activity areas. A 10-point Likert-type range was used to score the items (0= "I am not confident at all" and 100= "I am totally confident"). The overall average score is between 0 and 100. High scores will indicate a high level of physical activity efficacy.
The Physical Activity Questionnaire | Change from baseline to 8 weeks
  It will assess physical activity levels in children. It is is a self-administered, 7-day activity recall tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)